CLINICAL TRIAL: NCT05637554
Title: Laparoscopic Clipping Versus Extracorporeal Ligation in Complicated Appendicitis Upper Egypt Overview, Prospective Randomized Comparative Study
Brief Title: Laparoscopic Clipping Versus Extracorporeal Ligation in Complicated Appendicitis Upper Egypt Overview
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed Mohamed Elfoly, Resident Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laparoscopic appendectomy.
Record Dates: First submitted 2022-11-09; First posted 2022-12-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: Participants will be divided randomly into two groups, in the first group the investigators will use clipping in securing the base of the appendix but in other groups investigators will use extracorporeal ligation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic clipping appendectomy (Active Comparator): This group will undergo laparoscopic clipping of the base of the appendix during laparoscopic appendectomy.
  Interventions: Procedure: Laparoscopic appendectomy using clipping.
- Laparoscopic extracorporeal ligation appendectomy (Active Comparator): This group will undergo laparoscopic extracorporeal ligation of the base of the appendix during laparoscopic appendectomy.
  Interventions: Procedure: Laparoscopic appendectomy using extracorporeal ligation to secure the base of the appendix.

INTERVENTIONS:
Procedure: Laparoscopic appendectomy using clipping. — Laparoscopic appendectomy using clipping to secure the base of the appendix.
  Arms: Laparoscopic clipping appendectomy
Procedure: Laparoscopic appendectomy using extracorporeal ligation to secure the base of the appendix. — Laparoscopic appendectomy using extracorporeal ligation to secure the base of the appendix.
  Arms: Laparoscopic extracorporeal ligation appendectomy

SUMMARY:
The investigators aim to compare between laparoscopic clipping and extracorporeal ligation in complicated appendicitis regarding safety, efficacy, operative time, postoperative outcome, hospital stay and complications.

DETAILED DESCRIPTION:
Appendectomy has become one of the most commonly performed emergency abdominal operations since it's description by McBurney in the 1890s. Since laparoscopic appendectomy was first described in 1983, there is an increase in the general trend towards performing this surgery using laparoscopy instead of open technique as this approach shows better pain score, lesser use of analgesics, less operative complications, better post operative recovery, less hospital stay and rapid return to normal work.

There are many methods for securing the base of the appendix, some of which are expensive others are not available or technically demanding. In this study the investigators aim to compare between extracorporeal ligation and clipping techniques regarding feasibility, safety, efficacy, operative time, postoperative outcome and complications especially in complicated appendicitis.

AS management of complicated appendicitis laparoscopically is possible, secure and can lead to a little occurrence of infectious complications, fewer post-operative pain, quick revival and improve cosmesis so the investigators will do a prospective clinical trial comparative study between two common techniques to determine the best one in management of complicated cases.

ELIGIBILITY:
Inclusion Criteria:

* Acute complicated appendicitis.
* Perforated appendicitis (diagnosed intraoperatively)
* Patients who will undergo laparoscopic appendectomy.

Exclusion Criteria:

* Patients with straight forward appendectomy.
* Patients who are not fit for laparoscopic appendectomy.

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | After procedure completion, an average of 1 hour.
  Time of the total procedure.
Postoperative complications | Through study completion, an average of 1 year.
  All patients will be observed postoperatively for occurrence of complications as leakage, pelvic abscess, wound infection

SECONDARY OUTCOMES:
Hospital stay | Through the patient's hospital stay, an average of 1 week.
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Ali Riad Shaban, Professor, Principal Investigator — Assiut University; Moustafa Mahmoud Ebrahem, Principal Investigator — Assiut University; Moustafa Ali Sayed Mahmoud, Principal Investigator — Assiut University

REFERENCES:
- [Background] Bessoff KE, Choi J, Wolff CJ, Kashikar A, Carlos GM, Caddell L, Khan RI, Stave CD, Spain DA, Forrester JD. Evidence-based surgery for laparoscopic appendectomy: A stepwise systematic review. Surg Open Sci. 2021 Aug 26;6:29-39. doi: 10.1016/j.sopen.2021.08.001. eCollection 2021 Oct. PMID 34604728
- [Background] Casas MA, Dreifuss NH, Schlottmann F. High-volume center analysis and systematic review of stump appendicitis: solving the pending issue. Eur J Trauma Emerg Surg. 2022 Jun;48(3):1663-1672. doi: 10.1007/s00068-021-01707-y. Epub 2021 Jun 3. PMID 34085112
- [Background] Mannu GS, Sudul MK, Bettencourt-Silva JH, Cumber E, Li F, Clark AB, Loke YK. Closure methods of the appendix stump for complications during laparoscopic appendectomy. Cochrane Database Syst Rev. 2017 Nov 13;11(11):CD006437. doi: 10.1002/14651858.CD006437.pub3. PMID 29190038
- [Background] Delibegovic S, Mehmedovic Z. The influence of the different forms of appendix base closure on patient outcome in laparoscopic appendectomy: a randomized trial. Surg Endosc. 2018 May;32(5):2295-2299. doi: 10.1007/s00464-017-5924-z. Epub 2017 Nov 2. PMID 29098432